CLINICAL TRIAL: NCT04394936
Title: An Exploratory, Single-center, Double-blinded, Healthy Volunteer Controlled Study to Characterize Psoriasis Patients and Explore Novel Biomarkers for the Treatment Response of Psoriasis With a Multimodal Patient Profiling Approach.
Brief Title: An Explorative Psoriasis Biomarker Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early termination was initiated as the recruitment of the remaining 14 moderate-to-severe patients stagnated.
Sponsor: Centre for Human Drug Research, Netherlands (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHDR1806; 2019-002383-27 (EudraCT Number); NL70359.028.19 (Other: Regulatory registration number)
Record Dates: First submitted 2020-04-08; First posted 2020-05-20 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Psoriasis Vulgaris
Keywords: Psoriasis; Biomarker; Guselkumab
MeSH Terms: conditions — Psoriasis | interventions — guselkumab

STUDY DESIGN:
Intervention Model Description: This is an observational and interventional study in up to 40 patients with chronic plaque psoriasis and 10 healthy volunteers (observational only).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Guselkumab (Experimental): Guselkumab 100 mg/ml in prefilled syringe, subcutaneous injection, administered on day 0, 28 and 84.
  Interventions: Drug: Guselkumab
- Placebo (Placebo Comparator): Sodiumchloride 0,9% solution for injection, subcutaneous injection, administered on day 0, 28 and 84.
  Interventions: Drug: Placebos
- Healthy volunteers (No Intervention): Healthy volunteer cohort (observational)

INTERVENTIONS:
Drug: Guselkumab — 100 mg guselkumab administered subcutaneously
  Arms: Guselkumab
Drug: Placebos — Sodiumchloride 0,9% solution for injection
  Arms: Placebo

SUMMARY:
Plaque psoriasis may be an ideal model disease to explore potential therapeutic effects of immunosuppressive agents, given the easy accessibility of inflammatory lesions. In this study, the applicability of a systems dermatology approach is investigated in order to better assess the efficacy of psoriasis treatments at an early clinical stage. Up to this point, the clinical manifestation and regression of psoriasis is not yet sufficiently characterized with a multimodal state-of-the-art evaluation tool. The in-house developed 'DermaToolbox' enables the determination and subsequent integration of different diseaserelated biomarkers, including clinical, biophysical, molecular, cellular, and imaging markers as well as patient reported outcomes

DETAILED DESCRIPTION:
Psoriasis is a common skin disorder affecting up to an estimated 3% of the world's population. The most prevalent form of psoriasis, called psoriasis vulgaris or plaque psoriasis, is characterized by the presence of sharply demarcated erythematous plaques covered with white scales. These lesions can occur all over the body, but are most often seen on the extensor surface of the joints, nether regions and on the scalp. Patients can experience excessive itch, pain and sometimes bleeding of the lesions. Moreover, the visual appearance of psoriatic lesions can severely impact the patients psychological state and quality of life. An abundancy of different factors contributes to the pathogenesis of psoriasis. However, aberrant inflammatory reactions in the skin are thought to be the underlying cause. Excessive infiltration of immune cells in the skin and their interactions with cutaneous resident cells results in the hyper proliferation of keratinocytes and subsequent thickening of the epidermis. Indeed, more and more immunosuppressive biologicals targeting specific components of the immune system, like tumor necrosis factor alpha (TNFα), interleukin (IL-)17 and IL-23, have shown excellent efficacy in treating psoriasis Plaque psoriasis may be an ideal model disease to explore potential therapeutic effects of immunosuppressive agents, given the easy accessibility of inflammatory lesions and the good willingness of patients to participate in clinical studies. In this study, the applicability of a systems dermatology approach is investigated in order to better assess the efficacy of psoriasis treatments at an early clinical stage. Up to this point, the clinical manifestation and regression of psoriasis is not yet sufficiently characterized with a multimodal state-of-the-art evaluation tool. The in-house developed 'DermaToolbox' enables the determination and subsequent integration of different disease-related biomarkers, including clinical, biophysical, molecular, cellular, and imaging markers as well as patient-reported outcomes

ELIGIBILITY:
Inclusion Criteria Healthy volunteers

Eligible healthy volunteers must meet all of the following inclusion criteria at screening:

1. Male or non-pregnant female subjects, 18 to 75 years of age (inclusive);
2. Healthy as defined by the absence of any uncontrolled active or uncontrolled chronic disease following a medical and surgical history, documentation of general symptoms, and a symptom-directed physical examination including vital signs;
3. Willing to give written informed consent and willing and able to comply with the study protocol; Psoriasis patients

Eligible psoriasis patients must meet all of the following inclusion criteria at screening:

1. Male or non-pregnant female subjects, 18 to 75 years of age (inclusive);
2. Diagnosed with plaque psoriasis at least 6 months prior to study participation
3. Willing to discontinue any psoriasis therapy other than emollients.
4. Having mild (PASI ≥1 and ≤ 5) or moderate-to-severe (PASI ≥ 10) plaque psoriasis;
5. Currently not using psoriasis medication and ≥ 2 plaques suitable for repeated biopsies and target lesion assessments. At least one of these lesions must be located on the extremities, preferably on the elbow or knee, with a minimal target lesion score between 6 and 9. Or, when currently using psoriasis medication and insufficient lesional skin is present, willing to discontinue treatment awaiting rescreening (see also exclusion criteria 3 for psoriatic patients);
6. Willing to give written informed consent and willing and able to comply with the study protocol; Exclusion Criteria

Eligible healthy volunteers must meet none of the following exclusion criteria at screening:

1. History or symptoms of any uncontrolled, significant disease including (but not limited to), neurological, psychiatric, endocrine, cardiovascular, respiratory, gastrointestinal, hepatic, or renal disorder that may interfere with the study objectives, in the opinion of the Investigator;
2. History of immunological abnormality (e.g., immune suppression, severe allergy or anaphylaxis) that may interfere with study objectives, in the opinion of the Investigator;
3. Known infection requiring antibiotic therapy within the last three months prior to the study;
4. Immunosuppressive or immunomodulatory treatment within 30 days prior to the study;
5. Body mass index (BMI) ≤ 18.0 or ≥ 40.0 kg/m2;
6. Participation in an investigational drug study within 3 months prior to screening or more than 4 times a year;
7. Previous participation in an investigational drug study involving the dosing of an investigational compound targeting an immune pathway within one year prior to screening;
8. Loss or donation of blood over 500 mL within three months prior to screening;
9. The use of any medication or vitamin/mineral/herbal/dietary supplement within less than 5 half-lives prior to study participation, if the Investigator judges that it may interfere with the study objectives. The use of paracetamol (up to 4 g/day) is allowed;
10. History of alcohol consumption exceeding 5 standard drinks per day on average within 3 months of screening. Alcohol consumption will be prohibited from at least 12 hours preceding each study visit;
11. Any other condition that could interfere with the conduct of the study or the study objectives, in the opinion of the Investigator.

Psoriasis patients

Eligible psoriasis patients must meet none of the following exclusion criteria at screening:

1. Having primarily erythrodermic, pustular or guttate psoriasis;
2. Having medication-induced psoriasis;
3. Having previously failed on anti-IL23 therapy;
4. Having received treatments for psoriasis within the following intervals prior to the start of the study:

   1. < 2 weeks for topical treatment, e.g. retinoids, corticosteroids, vitamin D analogs
   2. < 4 weeks for phototherapy, e.g. PUVA, PDT
   3. < 4 weeks for non-biologic systemic treatment, e.g. retinoids, methotrexate, cyclosporine, fumaric acid esters
   4. < 4 weeks for etanercept
   5. < 8 weeks for adalimumab
   6. < 3 months for anti-IL17, anti-IL12(/23) and anti-IL23 treatments
5. History or symptoms of any significant uncontrolled disease including (but not limited to), neurological, psychiatric, endocrine, cardiovascular, respiratory, gastrointestinal, hepatic, or renal disorder that may interfere with the study objectives, in the opinion of the Investigator, excluding psoriasis and conditions that are related to psoriasis;
6. History of immunological abnormality (e.g., immune suppression, severe allergy or anaphylaxis) that may interfere with study objectives, in the opinion of the Investigator;
7. Known infection requiring antibiotic therapy within the last 3 months prior to the study, including latent tuberculosis;
8. Systemic immunosuppressive or immunomodulatory treatment within 30 days prior to the study;
9. Body mass index (BMI) ≤ 18.0 or ≥ 40.0 kg/m2;
10. Participation in an investigational drug study within 3 months prior to screening or more than 4 times a year;
11. Loss or donation of blood over 500 mL within three months prior to screening;
12. The use of any medication or vitamin/mineral/herbal/dietary supplement within less than 5 half-lives prior to study participation, if the Investigator judges that it may interfere with the study objectives. The use of paracetamol (up to 4 g/day) is allowed;
13. History of alcohol consumption exceeding 5 standard drinks per day on average within 3 months of screening. Alcohol consumption will be prohibited from at least 12 hours preceding each study visit;
14. Any other condition that could interfere with the conduct of the study or the study objectives, in the opinion of the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) Assessment | from day -14 to day 168
  Psoriasis Area and Severity Index (PASI) combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease).
Physicians Global Assesment (PGA) Assessment | from day -14 to day 168
  Physicians Global Assesment (PGA) is a 4-point scale ranging from 0 (no disease) to 4 (maximal disease).
Percentage body surface affected (%BSA) Assessment | from day -14 to day 168
  Percentage body surface affected (%BSA) is the area of lesional skin as a percentage of the total body surface
digital PASI | from day -14 to day 168
  Digital Psoriasis Area and Severity Index (dPASI) calculated from standardized total body photography
Erythema measurement of the skin | from day -14 to day 168
  Redness of the skin will be determined using a colorimeter
Multispectral imaging | from day -14 to day 168
  The redness and superficial morphology of (non-)lesional skin sites will be determined using a multispectral imaging system
Laser Speckle Contrast imaging | from day -14 to day 168
  The cutaneous microcirculation of (non-)lesional skin sites will be monitored over a 30 second timespan with a laser speckle contrast imager
Thermography | from day -14 to day 168
  Body surface temperature of (non-)lesional skin will be determined using a thermal imaging infrared camera
Patient reported outcomes | from day -14 to day 168
  Patients will be asked to report on their condition through an NRS scale (0 (better)- 10 (worse)) for sleeplessness, itch and quality of life. Additionally, patients image their lesions on a daily basis using a mobile device.
Activity Tracking Heartrate | from day -14 to day 168
  Subjects are requested to wear a smartwatch at all times which heart rate (beats per minute)
Activity Tracking Steps | from day -14 to day 168
  Subjects are requested to wear a smartwatch at all times which register steps (amount of steps taken)
Activity Tracking Sleep | from day -14 to day 168
  Subjects are requested to wear a smartwatch at all times which register sleep (hrs, minutes, seconds of rest)
Cells/ml; Circulating immune cell subsets | from day -14 to day 168
  Blood be drawn during using a venipuncture during visits and analyzed for the presence of immune cells (e.g. CD4+ and CD8+ T-Cells) using flow cytometry
Circulating protein biomarkers | from day -14 to day 168
  Blood be drawn during using a venipuncture during visits and analyzed for the presence of various chemokines and cytokines (e.g. CCL20, CCL17, CXCL8)
Anti-drug antibodies | from day 0 to day 168
  The occurrence of antibodies directed against guselkumab will be monitored during the treatment period (ng/ml)
Blister immune cell subsets | from day 0 to day 112
  Blisters will be induced on the non-lesional skin and the blister exudate aspirated. Blister exudate will be analyzed for the presence of immune cells (e.g. CD4+ and CD8+ T-Cells) using flow cytometry
Blister protein biomarkers | from day 0 to day 112
  Blisters will be induced on the non-lesional skin and blister fluid aspirated. Blister fluid will be analyzed for the presence of various chemokines and cytokines (e.g. CCL20, CCL17, CXCL8) (ng/ml)
Immunohistochemistry of biopsies | day 0 to day 112
  Biopsies will be sectioned and stained for the determination of the epidermal homeostasis (proliferation, differentiation and thickness) and infiltration of cellular immune subsets (e.g. presence of CD4 and CD8).
Transcriptome of biopsies | day 0 to day 112
  Biopsies will be analyzed with an untargeted next-generation sequencing approach.
Cutaneous microbiome | from day -14 to day 112
  The microbiome is collected by swabbing. The abundance of bacteria is thereafter determined using next-generation sequencing.
Fecal microbiome | from day 0 to day 112
  The bacterial composition of stool samples is determined using next-generation sequencing.
Skin surface biomarkers | from day -14 to day 112
  Superficial protein biomarkers are samples using a FibroTx Patch. Afterwards, these patches are extracted and the presence of protein biomarkers (e.g. HBD-3) determined using ELISA.
Lipidomics of the stratum corneum | from day -14 to day 112
  Tape stripping will be performed on (non-)lesional skin and lipids are subsequently extracted from the tape and analyzed using Liquid Chromatogrpahy-Mass Spectormetry. (ng/cm2)
Skin barrier function | from day -14 to day 168
  The trans epidermal water loss of (non-)lesional skin will be determined as function of the inside-out barrier function of the skin. (g/m2/h)
Patient genotyping | day -14
  A whole blood sample will be used to scan for common mutations in genes implicated in psoriasis using next-generation sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rissmann, PhD, Principal Investigator — Centre for Human Drug Research
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rousel J, Mergen C, Bergmans ME, Bruijnincx LJ, de Kam ML, Klarenbeek NB, Niemeyer-van der Kolk T, van Doorn MBA, Bouwstra JA, Rissmann R; Next-Generation ImmunoDermatology Consortium (NGID). Guselkumab treatment normalizes the stratum corneum ceramide profile and alleviates barrier dysfunction in psoriasis: results of a randomized controlled trial. J Lipid Res. 2024 Aug;65(8):100591. doi: 10.1016/j.jlr.2024.100591. Epub 2024 Jul 9. PMID 38992724